CLINICAL TRIAL: NCT00762788
Title: Clinical Trial of Several Contact Lenses in Extended Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CR-4472
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Investigator

ARMS (6):
- senofilcon A contact lens (Active Comparator): ACUVUE OASYS
  Interventions: Device: senofilcon A
- lotrafilcon A contact lens (Active Comparator): NIGHT&DAY
  Interventions: Device: lotrafilcon A
- lotrafilcon B contact lens (Active Comparator): O2Optix
  Interventions: Device: lotrafilcon B
- balafilcon A contact lens (Active Comparator): PureVision
  Interventions: Device: balafilcon A
- comfilcon A contact lens (Active Comparator): Biofinity
  Interventions: Device: comfilcon A
- etafilcon A contact lens (Active Comparator): ACUVUE 2
  Interventions: Device: etafilcon A

INTERVENTIONS:
Device: senofilcon A — 1 week extended wear contact lens
  Arms: senofilcon A contact lens
Device: lotrafilcon A — 1 week extended wear contact lens
  Arms: lotrafilcon A contact lens
Device: lotrafilcon B — 1 week extended wear contact lens
  Arms: lotrafilcon B contact lens
Device: balafilcon A — 1 week extended wear contact lens
  Arms: balafilcon A contact lens
Device: comfilcon A — 1 week extended wear contact lens
  Arms: comfilcon A contact lens
Device: etafilcon A — 1 week extended wear contact lens
  Arms: etafilcon A contact lens

SUMMARY:
The study is to clinically evaluate currently marketed contact lenses when used in an extended wear modality of up to seven days/six nights.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age, and be between 18 and 39 years of age.
* Signed Written Informed Consent and Investigator to record this on Case Report Form (CRF) in appropriate space.
* Require a visual correction in both eyes (Monovision not allowed)
* Require a soft contact lens spherical correction between -0.50 and -9.00D.
* Have an astigmatic correction less than 1.50D in both eyes.
* Be able to wear the lens powers available for this study.
* Be able to regularly wear the lenses on a 7 day/6 night extended wear basis (e.g. does not regularly swim more than once a week)
* Be correctable to a visual acuity of 20/30 or better in each eye.
* Have normal eyes with no evidence of abnormality or disease. For the purposes of this study a normal eye is defined as one having:
* No amblyopia.
* No evidence of lid abnormality or infection.
* No clinically significant slit lamp findings
* No other active ocular disease.
* No previous ocular surgery.

Exclusion Criteria:

* Requires concurrent ocular medication.
* Any systemic illness which would contraindicate lens wear or the medical treatment of which would affect vision or successful lens wear.
* No Clinically significant (Grade 3 or 4) slit lamp findings including corneal edema, corneal vascularization, corneal staining, tarsal abnormalities, bulbar injection, or any other abnormality of the cornea that would contraindicate contact lens wear.
* Diabetic.
* Infectious disease (e.g., hepatitis, tuberculosis) or an immunosuppressive disease (e.g., HIV).
* PMMA or RGP lens wear in the previous 8 weeks.
* Has had refractive surgery. Has had eye injury/surgery within 8 weeks immediately prior to enrolment for this study.
* Abnormal lacrimal secretions.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Keratoconus or other corneal irregularity.
* Pregnancy, lactating or planning a pregnancy at the time of enrollment only.
* Participation in any concurrent clinical trial.
* Currently wearing B&L PureVision, Ciba O2 Optix, Ciba Night & Day, CooperVision Biofinity, Vistakon ACUVUE® OASYS, or Vistakon ACUVUE®2 on an EW basis
* Has had previous adverse event(s) contraindicating EW e.g. MK or greater than 2 corneal scars which appear to be contact lens related (e.g. not trauma related).
* Has had an eye injury or surgery within the last eight weeks.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 2007-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vision Research Foundation, Chennai, Tamil Nadu, India

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 350 subjects recruited with 314 subjects being dispensed lenses. These 36 subjects were excluded due to failing to meet inclusion criteria.
Period: Overall Study
Arm/Group | Senofilcon A Contact Lens | Lotrafilcon A Contact Lens | Lotrafilcon B Contact Lens | Balafilcon A Contact Lens | Comfilcon A Contact Lens | Etafilcon A Contact Lens
Started | 55 | 58 | 42 | 64 | 43 | 52
Completed | 29 | 21 | 21 | 38 | 30 | 31
Not Completed | 26 | 37 | 21 | 26 | 13 | 21
Not completed — Lost to Follow-up | 26 | 37 | 21 | 26 | 13 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Senofilcon A Contact Lens | Lotrafilcon A Contact Lens | Lotrafilcon B Contact Lens | Balafilcon A Contact Lens | Comfilcon A Contact Lens | Etafilcon A Contact Lens | Total
Number analyzed (Participants) | 55 | 58 | 42 | 64 | 43 | 52 | 314
Age, Categorical [Count of Participants; unit: Participants] — Data was collected on those subjects 18 years and older, there were no pediatric patients enrolled in the study.
  Participants
    <=18 years | 11 | 13 | 11 | 15 | 7 | 12 | 69
    Between 18 and 65 years | 44 | 45 | 31 | 49 | 36 | 40 | 245
    >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.1 (3.2) | 21.6 (4.9) | 19.8 (1.7) | 21.0 (3.7) | 19.5 (1.3) | 20.6 (3.6) | 20.7 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 31 | 25 | 35 | 25 | 26 | 180
  Male | 17 | 27 | 17 | 29 | 18 | 26 | 134
Region of Enrollment [Number; unit: participants]
  India | 55 | 58 | 42 | 64 | 43 | 52 | 314

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Corneal Infiltrative Events
Description: Extended wear is defined as 7 days, 6 nights of lens wear, weekly replacement of lenses. Incidence was calculated as the number of subjects with event divided by the total number of subjects assigned to that lens type.
Time Frame: 52 weeks
Population: Subjects who were enrolled and dispensed lenses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Senofilcon A Contact Lens | Lotrafilcon A Contact Lens | Lotrafilcon B Contact Lens | Balafilcon A Contact Lens | Comfilcon A Contact Lens | Etafilcon A Contact Lens
Number analyzed (Participants) | 55 | 58 | 42 | 64 | 43 | 52
percentage of participants | 31 [20 to 44] | 16 [8 to 27] | 10 [4 to 22] | 8 [3 to 17] | 33 [20 to 47] | 10 [4 to 21]

2. Primary Outcome: Incidence of Adverse Events
Description: Occurrence of any Adverse Event by study lens. Incidence was calculated as the number of subjects with event divided by the total number of subjects assigned to that lens type.
Time Frame: 52 weeks
Population: Subjects who were enrolled and dispensed lenses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Senofilcon A Contact Lens | Lotrafilcon A Contact Lens | Lotrafilcon B Contact Lens | Balafilcon A Contact Lens | Comfilcon A Contact Lens | Etafilcon A Contact Lens
Number analyzed (Participants) | 55 | 58 | 42 | 64 | 43 | 52
percentage of participants | 35 [23 to 48] | 24 [15 to 37] | 19 [10 to 33] | 31 [21 to 43] | 37 [24 to 52] | 12 [5 to 23]

ADVERSE EVENTS:
Description: Significant Events were defined as events that are usually symptomatic and warrant either temporary or permanent discontinuation of lens wear. Non-significant Events were defined as events that are usually asymptomatic and do not warrant discontinuation of lens wear.
Arm/Group | Senofilcon A Contact Lens | Lotrafilcon A Contact Lens | Lotrafilcon B Contact Lens | Balafilcon A Contact Lens | Comfilcon A Contact Lens | Etafilcon A Contact Lens
Serious Adverse Events (participants affected / at risk) | 1/55 | 0/58 | 0/42 | 0/64 | 1/43 | 0/52
Other Adverse Events (participants affected / at risk) | 27/55 | 17/58 | 10/42 | 23/64 | 18/43 | 8/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Senofilcon A Contact Lens (N=55) | Lotrafilcon A Contact Lens (N=58) | Lotrafilcon B Contact Lens (N=42) | Balafilcon A Contact Lens (N=64) | Comfilcon A Contact Lens (N=43) | Etafilcon A Contact Lens (N=52)
Microbial Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Senofilcon A Contact Lens (N=55) | Lotrafilcon A Contact Lens (N=58) | Lotrafilcon B Contact Lens (N=42) | Balafilcon A Contact Lens (N=64) | Comfilcon A Contact Lens (N=43) | Etafilcon A Contact Lens (N=52)
CLPU (Eye disorders) | 7 (7) | 2 (2) | 1 (1) | 2 (2) | 8 (12) | 0 (0) — CLPU = Contact Lens Peripheral Ulcer; significant adverse event
SIE (Eye disorders) | 10 (11) | 5 (6) | 1 (1) | 3 (3) | 2 (2) | 5 (5) — SIE = Significant Infiltrative Event; significant adverse event
New Corneal Scar (Eye disorders) | 2 (2) | 3 (4) | 2 (3) | 0 (0) | 5 (5) | 0 (0) — New corneal scar without positive history; significant adverse events
Other Significant (Eye disorders) | 2 (2) | 2 (3) | 2 (2) | 3 (4) | 1 (1) | 0 (0) — Not specifically identified due to low counts of individual events
SLF Grade 2 or Less requiring Treatment (Eye disorders) | 1 (1) | 1 (1) | 3 (3) | 10 (12) | 2 (2) | 0 (0) — Slit lamp finding of Grade 1 or 2 (on 0-4 scale)
Other Non-significant (Eye disorders) | 5 (7) | 4 (6) | 1 (1) | 5 (6) | 0 (0) | 3 (6) — Not specifically identified due to low counts of individual events

LIMITATIONS AND CAVEATS:
Cautions for results: low completed enrollment numbers and number of non-neophytes lower than required per protocol. Arms not gender matched; Proportion of neophytes/non-neophytes not balanced; High rate of drop-out among subjects enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days